CLINICAL TRIAL: NCT04211363
Title: A Phase 3, 8-Week, Parallel Group, Double Blind, Vehicle-Controlled Study of the Safety and Efficacy of ARQ-151 Cream 0.3% Administered QD in Subjects With Chronic Plaque Psoriasis
Brief Title: Trial of PDE4 Inhibition With Roflumilast for the Management of Plaque Psoriasis
Acronym: DERMIS-1
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Arcutis Biotherapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: ARQ-151-301
Record Dates: First submitted 2019-12-23; First posted 2019-12-26 (Actual); Results first posted 2022-11-03 (Actual); Last update posted 2022-12-07 (Actual); Status verified 2022-12

CONDITIONS: Chronic Plaque Psoriasis
MeSH Terms: interventions — Roflumilast

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Rofumilast Cream 0.3% (Experimental): Participants receive roflumilast cream 0.3% once daily for 8 weeks.
  Interventions: Drug: Roflumilast 0.3% cream
- Vehicle cream (Placebo Comparator): Participants receive vehicle cream once daily for 8 weeks.
  Interventions: Drug: Vehicle Cream

INTERVENTIONS:
Drug: Roflumilast 0.3% cream — Roflumilast 0.3% cream for topical application.
  Other Names: ARQ-151
  Arms: Rofumilast Cream 0.3%
Drug: Vehicle Cream — Vehicle cream for topical application.
  Arms: Vehicle cream

SUMMARY:
This is a double-blind, parallel group, vehicle-controlled study to assess the safety and efficacy of roflumilast (ARQ-151) 0.3% cream vs vehicle (placebo) cream for treatment of chronic plaque psoriasis (CPP) in adult participants with 2 to 20% body surface area (BSA) of CPP.

ELIGIBILITY:
Inclusion Criteria:

* Participants legally competent to sign and give informed consent and if appropriate assent as required by local laws
* Males and females ages 2 years and older (inclusive)
* Clinical diagnosis of psoriasis vulgaris of at least 6 months duration (3 months for children) as determined by the Investigator
* Females of childbearing potential (FOCBP) must have a negative pregnancy test at Screening (Visit 1) and Baseline (Visit 2). In addition, sexually active FOCBP must agree to use at least one form of highly effective contraception throughout the trial.
* In good health as judged by the Investigator, based on medical history, physical examination, serum chemistry labs, hematology values, and urinalysis.
* Subjects considered reliable and capable of adhering to the Protocol and visit schedule, according to the judgment of the Investigator.

Exclusion Criteria:

* Planned excessive exposure of treated area(s) to either natural or artificial sunlight, tanning bed or other LED.
* Females who are pregnant, wishing to become pregnant during the study, or are breast-feeding.
* Previous treatment with ARQ-151 or its active ingredient
* Subjects with any serious medical condition or laboratory abnormality that would prevent study participation or place the subject at significant risk, as determined by the Investigator.
* Subjects with a history of chronic alcohol or drug abuse within 6 months of initiation of investigational product
* Subjects who are unable to communicate, read or understand the local language, or who display another condition, which in the Investigator's opinion, makes them unsuitable for clinical study participation

Min Age: 2 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 439 (Actual)
Dates: Start 2019-12-20 (Actual); Primary Completion 2020-11-16 (Actual); Study Completion 2020-11-16 (Actual)

CONTACTS AND LOCATIONS:
Locations (40):
- United States (31):
  - Arcutis Biotherapeutics Clinical Site 127, Encinitas, California
  - Arcutis Biotherapeutics Clinical Site 112, Fremont, California
  - Arcutis Biotherapeutics Clinical Site 120, Irvine, California
  - Arcutis Biotherapeutics Clinical Site 123, San Diego, California
  - Arcutis Biotherapeutics Clinical Site 136, San Francisco, California
  - Arcutis Biotherapeutics Clinical Site 118, Delray Beach, Florida
  - Arcutis Biotherapeutics Clinical Site 131, Miami, Florida
  - Arcutis Biotherapeutics Clinical Site 137, Ocala, Florida
  - Arcutis Biotherapeutics Clinical Site 105, Sanford, Florida
  - Arcutis Biotherapeutics Clinical Site 114, Plainfield, Illinois
  - Arcutis Biotherapeutics Clinical Site 102, Rolling Meadows, Illinois
  - Arcutis Biotherapeutics Clinical Site 111, Baton Rouge, Louisiana
  - Arcutis Biotherapeutics Clinical Site 125, Rockville, Maryland
  - Arcutis Biotherapeutics Clinical Site 138, Rockville, Maryland
  - Arcutis Biotherapeutics Clinical Site 101, Brighton, Massachusetts
  - Arcutis Biotherapeutics Clinical Site 116, Clinton Township, Michigan
  - Arcutis Biotherapeutics Clinical Site 139, Reno, Nevada
  - Arcutis Biotherapeutics Clinical Site 129, East Windsor, New Jersey
  - Arcutis Biotherapeutics Clinical Site 121, New York, New York
  - Arcutis Biotherapeutics Clinical Site 130, Rochester, New York
  - Arcutis Biotherapeutics Clinical Site 108, Stony Brook, New York
  - Arcutis Biotherapeutics Clinical Site 115, High Point, North Carolina
  - Arcutis Biotherapeutics Clinical Site 124, Fairborn, Ohio
  - Arcutis Biotherapeutics Clinical Site 134, Oklahoma City, Oklahoma
  - Arcutis Biotherapeutics Clinical Site 128, Duncansville, Pennsylvania
  - Arcutis Biotherapeutics Clinical Site 113, Exton, Pennsylvania
  - Arcutis Biotherapeutics Clinical Site 135, Pittsburgh, Pennsylvania
  - Arcutis Biotherapeutics Clinical Site 104, College Station, Texas
  - Arcutis Biotherapeutics Clinical Site 119, Dallas, Texas
  - Arcutis Biotherapeutics Clinical Site 110, San Antonio, Texas
  - Arcutis Biotherapeutics Clinical Site 117, San Antonio, Texas
- Canada (9):
  - Arcutis Biotherapeutics Clinical Site 132, Calgary, Alberta
  - Arcutis Biotherapeutics Clinical Site 103, London, Ontario
  - Arcutis Biotherapeutics Clinical Site 122, Markham, Ontario
  - Arcutis Biotherapeutics Clinical Site 133, Mississauga, Ontario
  - Arcutis Biotherapeutics Clinical Site 140, Ottawa, Ontario
  - Arcutis Biotherapeutics Clinical Site 109, Peterborough, Ontario
  - Arcutis Biotherapeutics Clinical Site 106, Waterloo, Ontario
  - Arcutis Biotherapeutics Clinical Site 107, Montreal, Quebec
  - Arcutis Biotherapeutics Clinical Site 126, Québec, Quebec

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Papp KA, Del Rosso JQ, Lebwohl MG, Gooderham MJ, Hebert AA, Hong HC, Kircik LH, Pariser DM, Stein Gold L, Strober B, Seal MS, Krupa D, Chu DH, Burnett P, Berk DR, Higham RC. Roflumilast Cream 0.3% in Patients with Chronic Plaque Psoriasis: Pooled PASI and PASI-HD Results from the DERMIS Phase III Trials. Dermatol Ther (Heidelb). 2025 Dec;15(12):3733-3744. doi: 10.1007/s13555-025-01562-4. Epub 2025 Oct 24. PMID 41134450
- [Derived] Thurston AW Jr, Osborne DW, Snyder S, Higham RC, Burnett P, Berk DR. Pharmacokinetics of Roflumilast Cream in Chronic Plaque Psoriasis: Data from Phase I to Phase III Studies. Am J Clin Dermatol. 2023 Mar;24(2):315-324. doi: 10.1007/s40257-022-00741-9. Epub 2022 Nov 24. PMID 36422852
- [Derived] Lebwohl MG, Kircik LH, Moore AY, Stein Gold L, Draelos ZD, Gooderham MJ, Papp KA, Bagel J, Bhatia N, Del Rosso JQ, Ferris LK, Green LJ, Hebert AA, Jones T, Kempers SE, Pariser DM, Yamauchi PS, Zirwas M, Albrecht L, Devani AR, Lomaga M, Feng A, Snyder S, Burnett P, Higham RC, Berk DR. Effect of Roflumilast Cream vs Vehicle Cream on Chronic Plaque Psoriasis: The DERMIS-1 and DERMIS-2 Randomized Clinical Trials. JAMA. 2022 Sep 20;328(11):1073-1084. doi: 10.1001/jama.2022.15632. PMID 36125472

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Adult male and female participants with chronic plaque psoriasis involving between 2% and 20% body surface area (BSA) [excluding the scalp, palms, and soles] were recruited at 43 study sites in the United States and Canada.
Groups:
- Rofumilast Cream 0.3%: Participants apply roflumilast cream 0.3% topically once daily for 8 weeks.
- Vehicle Cream: Participants apply vehicle cream topically once daily for 8 weeks.
Period: Overall Study
Arm/Group | Rofumilast Cream 0.3% | Vehicle Cream
Started | 286 | 153
Completed | 255 | 133
Not Completed | 31 | 20
Not completed — Adverse Event | 5 | 2
Not completed — Physician Decision | 0 | 1
Not completed — Protocol Violation | 1 | 0
Not completed — Pregnancy | 1 | 0
Not completed — Lost to Follow-up | 12 | 4
Not completed — Withdrawal by Subject | 11 | 11
Not completed — Other | 1 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Rofumilast Cream 0.3% | Vehicle Cream | Total
Number analyzed (Participants) | 286 | 153 | 439
Age, Continuous [Mean (Standard Deviation); unit: years] | 47.6 (14.09) | 48.7 (15.77) | 48.0 (14.69)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 97 | 57 | 154
  Male | 189 | 96 | 285
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 63 | 34 | 97
  Not Hispanic or Latino | 223 | 119 | 342
  Unknown or Not Reported | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 4 | 1 | 5
  Asian | 21 | 11 | 32
  Native Hawaiian or Other Pacific Islander | 2 | 0 | 2
  Black or African American | 8 | 8 | 16
  White | 234 | 124 | 358
  More than one race | 2 | 1 | 3
  Other | 15 | 8 | 23
Whole Body Investigator Global Assessment (IGA) Baseline Score [Count of Participants; unit: Participants] — The IGA is 5-point scale assessing the severity of plaque psoriasis, with scores ranging from 0 ('clear') to 4 ('severe'), with higher scores indicating greater plaque severity.
  Participants
    0 - Clear | 0 | 0 | 0
    1 - Almost Clear | 0 | 0 | 0
    2 - Mild | 51 | 20 | 71
    3 - Moderate | 206 | 122 | 328
    4 - Severe | 29 | 11 | 40
Intertriginous Area Investigator Global Assessment (I-IGA) Baseline Score [Count of Participants; unit: Participants] — For participants with intertriginous involvement, the I-IGA is 5-point scale assessing the severity of plaque psoriasis in the intertriginous area. Scores range from 0 ('clear') to 4 ('severe'), with higher scores indicating greater plaque severity. Population: Baseline I-IGA assessment was added in protocol amendment 1.
  Participants
    0 - Clear: number analyzed (Participants) | 68 | 33 | 101
    0 - Clear | 0 | 0 | 0
    1 - Almost Clear: number analyzed (Participants) | 68 | 33 | 101
    1 - Almost Clear | 5 | 1 | 6
    2 - Mild: number analyzed (Participants) | 68 | 33 | 101
    2 - Mild | 33 | 16 | 49
    3 - Moderate: number analyzed (Participants) | 68 | 33 | 101
    3 - Moderate | 27 | 16 | 43
    4 - Severe: number analyzed (Participants) | 68 | 33 | 101
    4 - Severe | 3 | 0 | 3
Baseline Psoriasis Symptom Diary (PSD) Total Baseline Score [Mean (Standard Deviation); unit: score on a scale] — The PSD is a 16-item questionnaire asking subjects to rate the severity of psoriasis-related symptoms in the past 24 hours. Each question is scored from 0 ("no symptoms") to 10 ("worst imaginable symptoms"). Scores range from 0 to 160, with higher scores indicating greater symptom severity. Population: All participants with baseline PSD total scores available are included.
  score on a scale
    number analyzed (Participants) | 282 | 150 | 432
    (all) | 72.1 (42.75) | 73.4 (41.29) | 72.6 (42.21)
Worst Itch Numerical Rating Scale (WI-NRS) Baseline Score [Count of Participants; unit: Participants] — The WI-NRS is a simple, single item scale to assess the subject-reported severity of this symptom, on a scale ranging from 0 ("no itch") to 10 ("worst imaginable itch") the subject experienced in the previous 24 hours. Higher scores indicate greater symptom severity. Population: One participant in the Roflumilast Cream 0.3% arm did not have a baseline WI-NRS assessment.
  Participants
    0: number analyzed (Participants) | 285 | 153 | 438
    0 | 16 | 12 | 28
    1: number analyzed (Participants) | 285 | 153 | 438
    1 | 11 | 5 | 16
    2: number analyzed (Participants) | 285 | 153 | 438
    2 | 14 | 11 | 25
    3: number analyzed (Participants) | 285 | 153 | 438
    3 | 26 | 10 | 36
    4: number analyzed (Participants) | 285 | 153 | 438
    4 | 26 | 7 | 33
    5: number analyzed (Participants) | 285 | 153 | 438
    5 | 32 | 14 | 46
    6: number analyzed (Participants) | 285 | 153 | 438
    6 | 37 | 26 | 63
    7: number analyzed (Participants) | 285 | 153 | 438
    7 | 34 | 20 | 54
    8: number analyzed (Participants) | 285 | 153 | 438
    8 | 49 | 23 | 72
    9: number analyzed (Participants) | 285 | 153 | 438
    9 | 20 | 19 | 39
    10: number analyzed (Participants) | 285 | 153 | 438
    10 | 20 | 6 | 26

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Achieving Success in Investigator Global Assessment (IGA) Scale Assessment of Disease Severity at Week 8
Description: The number of participants achieving "success" in IGA assessment of disease severity at Week 8 is presented (observed data only) for each arm. Success was defined as achievement of an IGA score of 0 ('clear') or 1 ('almost clear') at Week 8, accompanied by a ≥2-grade improvement from baseline IGA score. The IGA is a 5-point scale assessing the severity of plaque psoriasis, with scores ranging from 0 ('clear') to 4 ('severe'), and higher scores indicate greater symptom severity.
Time Frame: Baseline (Day 1) and Week 8
Population: All randomized participants with data available are included.
Measure: Count of Participants; unit: Participants
Arm/Group | Rofumilast Cream 0.3% | Vehicle Cream
Number analyzed (Participants) | 255 | 132
Participants | 108 | 8
Statistical Analysis 1: Comparison: Rofumilast Cream 0.3% vs Vehicle Cream; IGA Success Odds Ratio; Test type: Superiority; p < 0.0001, Cochran-Mantel-Haenszel; Stratified by pooled study site, baseline IGA, and baseline intertriginous involvement per randomization with multiple imputation of missing data; Odds Ratio (OR) = 20.69, 95% CI 2-sided [7.58 to 56.48] — Common odds ratio stratified by pooled study site, baseline IGA, and baseline intertriginous involvement per randomization with multiple imputation of missing data

2. Secondary Outcome: Time to Achieve Psoriasis Area Severity Index-50 (PASI-50)
Description: The Psoriasis Area and Severity Index (PASI) is widely used for the measurement of severity of psoriasis. PASI combines the assessment of the severity of lesions and the area affected into a single score in the range from 0 (no disease) to 72 (maximal disease), with higher scores indicating greater symptom severity. The time to achieve PASI-50 (defined as a 50% reduction from baseline in PASI score) is presented, and is based on observed data only.
Time Frame: From start of treatment to achievement of PASI-50 or study completion/early termination (maximum duration = 121 days)
Population: All randomized participants are included.
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Rofumilast Cream 0.3% | Vehicle Cream
Number analyzed (Participants) | 286 | 153
days | 31.0 [29.0 to 41.0] | 104.0 [85.0 to NA] — Upper bound of 95% CI was not estimable due to low number of cases.
Statistical Analysis 1: Comparison: Rofumilast Cream 0.3% vs Vehicle Cream; Time to PASI-50; Test type: Superiority; p < 0.0001, Log Rank; Unstratified log-rank test; Hazard Ratio (HR) = 3.867, 95% CI 2-sided [2.795 to 5.351] — Stratified by pooled study site, baseline IGA, and baseline intertriginous involvement per randomization

3. Secondary Outcome: Number of Participants Achieving Psoriasis Area Severity Index 75 (PASI-75)
Description: The Psoriasis Area and Severity Index (PASI) is widely used for the measurement of severity of psoriasis. PASI combines the assessment of the severity of lesions and the area affected into a single score in the range from 0 (no disease) to 72 (maximal disease), with higher scores indicating greater symptom severity. The number of participants achieving PASI-75 (defined as a 75% reduction from baseline in PASI score) at Week 8 is presented. Participant counts are based on observed data only.
Time Frame: Baseline (Day 1) and Week 8
Population: All randomized participants with data available at Week 8 are included.
Measure: Count of Participants; unit: Participants
Arm/Group | Rofumilast Cream 0.3% | Vehicle Cream
Number analyzed (Participants) | 255 | 132
Participants | 106 | 10
Statistical Analysis 1: Comparison: Rofumilast Cream 0.3% vs Vehicle Cream; PASI-75 at Week 8 Odds Ratio; Test type: Superiority; p < 0.0001, Cochran-Mantel-Haenszel; [statistical method as in outcome 1, analysis 1]; Odds Ratio (OR) = 12.00, 95% CI 2-sided [5.15 to 27.93] — [estimate comment as in outcome 1, analysis 1]

4. Secondary Outcome: Number of Participants Achieving Psoriasis Area Severity Index-90 (PASI-90)
Description: Psoriasis Area and Severity Index (PASI) is widely used for the measurement of severity of psoriasis. PASI combines the assessment of the severity of lesions and the area affected into a single score in the range 0 (no disease) to 72 (maximal disease) [higher scores indicate greater symptom severity]. The number of participants achieving PASI-90 (defined as a 90% reduction from baseline in PASI score) at Week 8 is presented. Participant counts are based on observed data only.
Time Frame: Baseline (Day 1) and Week 8
Population: All randomized participants with data available at Week 8 are included.
Measure: Count of Participants; unit: Participants
Arm/Group | Rofumilast Cream 0.3% | Vehicle Cream
Number analyzed (Participants) | 255 | 132
Participants | 57 | 3
Statistical Analysis 1: Comparison: Rofumilast Cream 0.3% vs Vehicle Cream; PASI-90 at Week 8 Odds Ratio; Test type: Superiority; p < 0.0001, Cochran-Mantel-Haenszel; Stratified by study site, baseline IGA score, and baseline intertriginous involvement with multiple imputation of missing data; Odds Ratio (OR) = 17.90, 95% CI 2-sided [4.38 to 73.09] — Cochran-Mantel-Haenszel stratified by study site, baseline IGA score, and baseline intertriginous involvement with multiple imputation of missing data

5. Secondary Outcome: Number of Participants Achieving Intertriginous IGA (I-IGA) Success at Week 8
Description: The number of participants achieving I-IGA success at Week 8 is presented. Success is defined as achievement of I-IGA score of 0 ('clear') or 1 ('almost clear') at Week 8 PLUS a ≥2-grade improvement in score from Baseline. The I-IGA is a 5-point scale assessing the severity of plaque psoriasis in the intertriginous area, with scores ranging from 0 ('clear') to 4 ('severe'), with higher scores indicating greater symptom severity. Participant counts are based on observed data only.
Time Frame: Baseline (Day 1) and Week 8
Population: All randomized participants with intertriginous area involvement an I-IGA score at Baseline ≥ 2 and who have Week 8 data available are included.
Measure: Count of Participants; unit: Participants
Arm/Group | Rofumilast Cream 0.3% | Vehicle Cream
Number analyzed (Participants) | 52 | 29
Participants | 37 | 4
Statistical Analysis 1: Comparison: Rofumilast Cream 0.3% vs Vehicle Cream; I-IGA Success at Week 8 Odds Ratio; Test type: Superiority; p < 0.0001, Cochran-Mantel-Haenszel; Stratified by pooled study site and baseline IGA per randomization with multiple imputation of missing data; Odds Ratio (OR) = 17.94, 95% CI 2-sided [2.33 to 138.20] — Common odds ratio stratified by pooled study site and baseline IGA per randomization with multiple imputation of missing data

6. Secondary Outcome: Number of Participants Achieving Score of 'Clear' in I-IGA at Week 8
Description: The number of participants achieving an IGA score of 0 ('clear') at Week 8 is presented (observed data only) for each arm. The I-IGA is a 5-point scale assessing the severity of plaque psoriasis, with scores ranging from 0 ('clear') to 4 ('severe'); higher scores indicate greater symptom severity.
Time Frame: Week 8
Population: as for outcome 5
Measure: Count of Participants; unit: Participants
Arm/Group | Rofumilast Cream 0.3% | Vehicle Cream
Number analyzed (Participants) | 52 | 29
Participants | 33 | 3
Statistical Analysis 1: Comparison: Rofumilast Cream 0.3% vs Vehicle Cream; I-IGA Clear at Week 8 Odds Ratio; Test type: Superiority; p = 0.003, Cochran-Mantel-Haenszel; Stratified by pooled study site and baseline IGA per randomization with multiple imputation of missing data; Odds Ratio (OR) = 29.36, 95% CI 2-sided [2.99 to 288.36] — [estimate comment as in outcome 5, analysis 1]

7. Secondary Outcome: Number of Participants Achieving Worst Itch Numerical Rating Score (WI-NRS) Success
Description: The number of participants achieving success in WI-NRS is presented. Success is defined as achievement of a ≥ 4-point reduction in WI-NRS pruritus score in participants with WI-NRS pruritus score ≥ 4 at baseline. The WI-NRS is a 10 point scale ranging from 0 ('no itch') to 10 ('worst itch imaginable'), with higher scores indicating greater symptoms severity. Results are based on observed data only.
Time Frame: Baseline (Day 1) and Weeks 2, 4, and 8
Population: All randomized participants with WI-NRS pruritus score ≥4 at baseline and data available at the relevant time points are included.
Measure: Count of Participants; unit: Participants
Arm/Group | Rofumilast Cream 0.3% | Vehicle Cream
Number analyzed (Participants) | 218 | 115
Participants
  Week 2 Observed Data: number analyzed (Participants) | 209 | 109
  Week 2 Observed Data | 73 | 24
  Week 4 Observed Data: number analyzed (Participants) | 201 | 100
  Week 4 Observed Data | 101 | 18
  Week 8 Observed Data: number analyzed (Participants) | 191 | 97
  Week 8 Observed Data | 129 | 26
Statistical Analysis 1: Comparison: Rofumilast Cream 0.3% vs Vehicle Cream; WI-NRS Success at Week 2 Odds Ratio; Test type: Superiority; p = 0.1197, Cochran-Mantel-Haenszel; [statistical method as in outcome 1, analysis 1]; Odds Ratio (OR) = 1.76, 95% CI 2-sided [0.98 to 3.19] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Rofumilast Cream 0.3% vs Vehicle Cream; WI-NRS Success at Week 4 Odds Ratio; Test type: Superiority; p < 0.0001, Cochran-Mantel-Haenszel; [statistical method as in outcome 1, analysis 1]; Odds Ratio (OR) = 4.36, 95% CI 2-sided [2.31 to 8.26] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 3: Comparison: Rofumilast Cream 0.3% vs Vehicle Cream; WI-NRS at Week 8 Odds Ratio; Test type: Superiority; p < 0.0001, Cochran-Mantel-Haenszel; [statistical method as in outcome 1, analysis 1]; Odds Ratio (OR) = 7.84, 95% CI 2-sided [3.85 to 15.94] — [estimate comment as in outcome 1, analysis 1]

8. Secondary Outcome: Change From Baseline in Psoriasis Symptoms Diary (PSD) Score
Description: The PSD is a 16-item questionnaire asking subjects to rate the severity of psoriasis-related symptoms in the past 24 hours. Each question is scored from 0 ("no symptoms") to 10 ("worst imaginable symptoms"). Scores range from 0 to 160, with higher scores indicating greater symptom severity. The least squares (LS) mean (95% CI) change in PSD total score relative to baseline is presented for each treatment arm, with decreases from baseline indicating symptom improvement.
Time Frame: Weeks 4 and 8
Population: All randomized participants are included.
Measure: Least Squares Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Rofumilast Cream 0.3% | Vehicle Cream
Number analyzed (Participants) | 286 | 153
score on a scale
  Week 4 | -43.5 [-48.2 to -38.9] | -17.7 [-23.5 to -11.9]
  Week 8 | -50.1 [-55.0 to -45.1] | -19.2 [-25.3 to -13.0]
Statistical Analysis 1: Comparison: Rofumilast Cream 0.3% vs Vehicle Cream; Comparison of change from baseline in PSD score at Week 4; Test type: Superiority; p < 0.0001, ANCOVA; Site, baseline IGA, baseline intertriginous involvement, and baseline PSD scores were independent variables, multiple imputation used for missing data; Mean Difference (Final Values) = -25.83, 95% CI 2-sided [-31.7 to -20.0] — Site, baseline IGA, baseline intertriginous involvement, and baseline PSD scores were independent variables, multiple imputation used for missing data
Statistical Analysis 2: Comparison: Rofumilast Cream 0.3% vs Vehicle Cream; Comparison of change from baseline in PSD score at Week 8; Test type: Superiority; p < 0.0001, ANCOVA; [statistical method as in outcome 8, analysis 1]; Mean Difference (Final Values) = -30.9, 95% CI 2-sided [-37.2 to -24.6] — [estimate comment as in outcome 8, analysis 1]

ADVERSE EVENTS:
Time Frame: Up to 121 days
Description: All participants who received ≥1 dose of study drug are included.
Arm/Group | Rofumilast Cream 0.3% | Vehicle Cream
All-Cause Mortality (participants affected / at risk) | 0/286 | 0/153
Serious Adverse Events (participants affected / at risk) | 2/286 | 1/153
Other Adverse Events (participants affected / at risk) | 0/286 | 0/153
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Rofumilast Cream 0.3% (N=286) | Vehicle Cream (N=153)
Concussion (Injury, poisoning and procedural complications) | 1 | 0
Foot fracture (Injury, poisoning and procedural complications) | 1 | 0
Deformity thorax (Musculoskeletal and connective tissue disorders) | 1 | 0
Plasma cell myeloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Sponsor is supportive of publishing clinical trial findings. The process of coordinating publication efforts is detailed in the Clinical Trial Agreement.

DOCUMENTS (2):
  • Study Protocol (2020-02-21): https://cdn.clinicaltrials.gov/large-docs/63/NCT04211363/Prot_000.pdf
  • Statistical Analysis Plan (2020-12-16): https://cdn.clinicaltrials.gov/large-docs/63/NCT04211363/SAP_001.pdf